CLINICAL TRIAL: NCT00988884
Title: A Phase III Open-Label Clinical Trial to Study the Immunogenicity and Tolerability of V503 (A Multivalent Human Papillomavirus [HPV] L1 Virus-Like Particle [VLP] Vaccine) Given Concomitantly With Menactra™ and Adacel™ in Preadolescents and Adolescents (11 to 15 Year Olds)
Brief Title: A Study of V503 Given Concomitantly With Menactra™ and Adacel™ in 11 to 15 Year Olds (V503-005)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V503-005; V503-005
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-11

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Concomitant Vaccination (Experimental): V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm on Day 1, Month 2, and Month 6, and Menactra™ and Adacel™ each given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm on Day 1
  Interventions: Biological: V503; Biological: Comparator: Menactra™ (Concomitant); Biological: Comparator: Adacel™ (Concomitant)
- Non-concomitant Vaccination (Experimental): V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm on Day 1, Month 2, and Month 6, and Menactra™ and Adacel™ each given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Month 1
  Interventions: Biological: V503; Biological: Comparator: Menactra™ (Non-Concomitant); Biological: Comparator: Adacel™ (Non-concomitant)

INTERVENTIONS:
Biological: V503 — V503 (Multivalent HPV L1 VLP vaccine) given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm at Day 1, Month 2, and Month 6
Biological: Comparator: Menactra™ (Concomitant) — Menactra™ given as a single 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm on Day 1.
  Arms: Concomitant Vaccination
Biological: Comparator: Adacel™ (Concomitant) — Adacel™ given as a single 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm on Day 1.
  Arms: Concomitant Vaccination
Biological: Comparator: Menactra™ (Non-Concomitant) — Menactra™ given as a single 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Month 1.
  Arms: Non-concomitant Vaccination
Biological: Comparator: Adacel™ (Non-concomitant) — Adacel™ given as a single 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Month 1.
  Arms: Non-concomitant Vaccination

SUMMARY:
This study will evaluate the tolerability and immunogenicity of administration of the first dose of V503 at the same time as Menactra™ and Adacel™ versus administration of V503 one month prior to administration of Menactra™ and Adacel™.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject's parent/legal guardian can read, understand, and complete the vaccine report card
* Subject is not sexually active and does not plan on becoming sexually active during the study
* Subject has received a documented full primary immunization series against diphtheria, tetanus, and pertussis (not in the last 5 years)

Exclusion Criteria:

* Subject has a known allergy to any vaccine component of V503, Menactra™, or Adacel™
* Subject has a condition that is a contraindication to vaccination with Menactra™ or Adacel™
* Subject has any coagulation disorder
* Female subject is pregnant
* Subject is immunocompromised or immunodeficient
* Subject has had a splenectomy
* Subject has received immunosuppressive therapies in the prior year
* Subject has received any immune globulin product or blood-derived product in the last 3 months
* Subject has received inactivated vaccines within 14 days or live vaccines within 21 days of the first study vaccination
* Subject has received a marketed HPV vaccine or has participation in an HPV vaccine trial
* Subject has received a meningococcal vaccine
* Subject has a fever >= 100F within 24 hours of vaccination
* Subject has a history of HPV

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1241 (Actual)
Dates: Start 2009-10-21 (Actual); Primary Completion 2011-02-22 (Actual); Study Completion 2011-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rodrigues S, Grenha A. Activation of Macrophages: Establishing a Role for Polysaccharides in Drug Delivery Strategies Envisaging Antibacterial Therapy. Curr Pharm Des. 2015;21(33):4869-87. doi: 10.2174/1381612821666150820103910. PMID 26290207
- [Result] Schilling A, Parra MM, Gutierrez M, Restrepo J, Ucros S, Herrera T, Engel E, Huicho L, Shew M, Maansson R, Caldwell N, Luxembourg A, Ter Meulen AS. Coadministration of a 9-Valent Human Papillomavirus Vaccine With Meningococcal and Tdap Vaccines. Pediatrics. 2015 Sep;136(3):e563-72. doi: 10.1542/peds.2014-4199. Epub 2015 Aug 3. PMID 26240207
- [Result] Moreira ED Jr, Block SL, Ferris D, Giuliano AR, Iversen OE, Joura EA, Kosalaraksa P, Schilling A, Van Damme P, Bornstein J, Bosch FX, Pils S, Cuzick J, Garland SM, Huh W, Kjaer SK, Qi H, Hyatt D, Martin J, Moeller E, Ritter M, Baudin M, Luxembourg A. Safety Profile of the 9-Valent HPV Vaccine: A Combined Analysis of 7 Phase III Clinical Trials. Pediatrics. 2016 Aug;138(2):e20154387. doi: 10.1542/peds.2015-4387. Epub 2016 Jul 15. PMID 27422279
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=V503-005&kw=V503-005&tab=access

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-concomitant Vaccination: V503 given as a 0.5 mL intramuscular injection in the deltoid muscle of the non-dominant arm at Day 1, Month 2, and Month 6, and Menactra™ and Adacel™ each given as a 0.5 mL intramuscular injection in the deltoid muscle of the dominant arm at Month 1
Period: Overall Study
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Started | 621 | 620
Completed | 586 | 584
Not Completed | 35 | 36
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 20 | 16
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 15 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination | Total
Number analyzed (Participants) | 621 | 620 | 1241
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.2 (1.4) | 12.1 (1.3) | 12.2 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 310 | 621
  Male | 310 | 310 | 620

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of the Antibody Response to Each of the Human Papillomavirus (HPV) Types Contained in V503
Description: Serum antibody titers to HPV Types 6, 11, 16, 18, 31, 33, 45, 52, and 58 were evaluated using a competitive Luminex immunoassay. Titers are reported in milli Merck Units/mL.
Time Frame: 4 weeks following Month 6 vaccination
Population: The per-protocol population included participants who received all study vaccinations, were seronegative to HPV on Day 1, and had serum samples available for evaluation of the endpoint
Measure: Geometric Mean (Full Range); unit: milli Merck Units/mL
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
milli Merck Units/mL
  Anti-HPV 6: n=501, 514 | 2198.7 [137.0 to 18555.0] | 2260.7 [210.0 to 30594.0]
  Anti-HPV 11: n=502, 514 | 1495.0 [64.0 to 13292.0] | 1547.2 [109.0 to 30345.0]
  Anti-HPV 16: n=513, 530 | 8882.6 [159.0 to 60653.0] | 9027.6 [619.0 to 125497.0]
  Anti-HPV 18: n=516, 535 | 2610.4 [35.0 to 49077.0] | 2633.9 [79.0 to 45639.0]
  Anti-HPV 31: n=514, 536 | 2439.4 [50.0 to 43734.0] | 2334.3 [89.0 to 45636.0]
  Anti-HPV 33: n=520, 537 | 1268.5 [25.0 to 34514.0] | 1276.3 [52.0 to 21991.0]
  Anti-HPV 45: n=523, 539 | 947.8 [8.0 to 15268.0] | 863.8 [16.0 to 13822.0]
  Anti-HPV 52: n=521, 538 | 1082.7 [26.0 to 10420.0] | 1103.7 [50.0 to 20926.0]
  Anti-HPV 58: n=519, 537 | 1532.8 [32.0 to 14833.0] | 1555.1 [46.0 to 32108.0]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 6; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 95% confidence interval for the fold difference is >0.5; p < 0.001, ANOVA; Fold difference in GMT = 0.97, 95% CI 2-sided [0.88 to 1.08]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 11; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.97, 95% CI 2-sided [0.87 to 1.07]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 16; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.98, 95% CI 2-sided [0.89 to 1.09]
Statistical Analysis 4: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 18; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.99, 95% CI 2-sided [0.88 to 1.12]
Statistical Analysis 5: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 31; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 1.04, 95% CI 2-sided [0.93 to 1.17]
Statistical Analysis 6: Comparison: Concomitant Vaccination; Anti-HPV 33; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.99, 95% CI 2-sided [0.89 to 1.11]
Statistical Analysis 7: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 45; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 1.10, 95% CI 2-sided [0.97 to 1.25]
Statistical Analysis 8: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 52; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.98, 95% CI 2-sided [0.88 to 1.10]
Statistical Analysis 9: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-HPV 58; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.99, 95% CI 2-sided [0.88 to 1.10]

2. Primary Outcome: Percentage of Participants With >=4-fold Increase in Antibody Titers to Neisseria Meningitidis Serogroups
Description: For the Concomitant Vaccination group, serum samples were collected at Day 1 (baseline) and 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected at Month 1 (baseline) and 4 weeks after the Month 1 vaccination. Bactericidal antibodies to Neisseria meningitidis serogroups A, C, Y, and W-135 were measured by incubating serial dilutions of serum with target N. meningitidis strains and complement, and enumerating the surviving bacteria after overnight incubation on blood agar plates. The serum bactericidal titer is reported as the reciprocal of the final serum dilution giving >50% killing in 60 minutes.
Time Frame: Baseline and 4 weeks following Day 1 (Concomitant) or Month 1 (Non-concomitant) vaccination
Population: The per-protocol population included participants who received study vaccination and had serum samples available for evaluation of the endpoint
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
Percentage of participants
  Serogroup A: n=590, 564 | 79.0 | 75.4
  Serogroup C:n=590, 566 | 92.9 | 95.1
  Serogroup Y: n=590, 566 | 91.5 | 89.4
  Serogroup W-135: n=589, 566 | 95.6 | 97.7
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Serogroup A; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 97.5% confidence interval for the percentage difference is greater than -10; p < 0.001, Miettinen and Nurminen; Difference in percentage = 3.8, 97.5% CI 2-sided [-1.7 to 9.3]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Serogroup C; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = -2.1, 97.5% CI 2-sided [-5.4 to 1.1]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Serogroup Y; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 2.1, 97.5% CI 2-sided [-1.8 to 6.1]
Statistical Analysis 4: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Serogroup W-135; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = -2.1, 97.5% CI 2-sided [-4.7 to 0.3]

3. Primary Outcome: Percentage of Participants Who Achieve Acceptable Titers of Anti-Diphtheria and Anti-Tetanus Antibody
Description: For the Concomitant Vaccination group, serum samples were collected 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after the Month 1 vaccination. Titers of neutralizing antibody to diphtheria toxin were measured using a cell-based Diphtheria Micrometabolic Inhibition assay. The lower limit of quantitation of the assay was defined as 0.01 International Units (IU)/mL. Serum titers of neutralizing antibody to tetanus toxin were measured using an enzyme immunoassay. The lower limit of quantitation of the assay was defined as 0.04 IU/mL. Acceptable titers refer to the World Health Organization-defined protective titers of >=0.1 IU/mL.
Time Frame: 4 weeks following Day 1 or Month 1 vaccination
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
Percentage of participants
  Anti-diphtheria titer >=0.1 IU/mL: n=595, 566 | 100 | 100
  Anti-tetanus titer >=0.1 IU/mL: n=594, 562 | 99.8 | 100
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-diphtheria titer >=0.1 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = 0.0, 97.5% CI 2-sided [-0.8 to 0.9]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-tetanus titer >=0.1 IU/mL; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in percentage = -0.2, 97.5% CI 2-sided [-1.2 to 0.7]

4. Primary Outcome: Geometric Mean Titers of Pertussis Antibody Responses
Description: For the Concomitant Vaccination group, serum samples were collected 4 weeks after the Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after the Month 1 vaccination. Titers of anti-pertussis toxin (PT), anti-filamentous hemagglutinin (FHA), anti-pertactin (PRN), and anti-fimbriae 2/3 (FM 2/3) antibodies were measured using enzyme-linked immunosorbent assays. The titers were expressed as Enzyme-linked Immunoassay Units (ELU)/mL.
Time Frame: 4 weeks following Day 1 or Month 1 vaccination
Population: as for outcome 2
Measure: Geometric Mean (Full Range); unit: ELU/mL
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
ELU/mL
  Anti-PT: n=595, 566 | 28.5 [2.5 to 1056.0] | 35.7 [2.5 to 618.0]
  Anti-FHA: n=595, 566 | 184.1 [5.0 to 3019.0] | 201.4 [3.0 to 1547.0]
  Anti-PRN: n=595, 566 | 328.4 [15.0 to 5093.0] | 344.0 [19.0 to 3232.0]
  Anti-FIM 2/3: n=595, 566 | 653.0 [2.5 to 73900.0] | 681.4 [2.5 to 27520.0]
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-PT; Test type: Non-Inferiority or Equivalence — Noninferiority of concomitant versus non-concomitant vaccination is demonstrated if the lower limit of the 97.5% confidence interval for the fold difference is >0.67; p = 0.003, ANOVA; Fold difference in GMT = 0.80, 97.5% CI 2-sided [0.69 to 0.92]
Statistical Analysis 2: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-FHA; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.91, 97.5% CI 2-sided [0.83 to 1.01]
Statistical Analysis 3: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-PRN; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.95, 97.5% CI 2-sided [0.84 to 1.08]
Statistical Analysis 4: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Anti-FIM 2/3; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; p < 0.001, ANOVA; Fold difference in GMT = 0.96, 97.5% CI 2-sided [0.76 to 1.21]

5. Primary Outcome: Percentage of Participants With a V503 Injection-site Adverse Experience
Description: An adverse experience (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Only injection-site AEs in the arm that received V503 vaccination were reported for this endpoint.
Time Frame: Day 1 through Day 5 following Day 1 vaccination
Population: The population analyzed included all vaccinated participants with follow-up for injection-site AEs
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 611 | 609
Percentage of participants | 59.9 | 58.0

6. Primary Outcome: Percentage of Participants With a Menactra™ or Adacel™ Injection-site Adverse Experience
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study vaccine, whether or not considered related to the use of the vaccine. Any worsening of a preexisting condition which is temporally associated with the use of the study vaccine is also an AE. Only injection-site AEs in the arm that received Menactra™ and Adacel™ vaccination were reported for this endpoint. For the Concomitant Vaccination group, injection-site AEs are reported following Day 1 vaccination; for the Non-concomitant Vaccination group, injection-site AEs are reported following Month 1 vaccination.
Time Frame: Day 1 through Day 5 following Day 1 or Month 1 vaccination
Population: The population analyzed included all vaccinated participants with follow-up for injection-site AEs
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 611 | 598
Percentage of participants | 74.6 | 70.7

7. Primary Outcome: Percentage of Participants With Maximum Temperature >=37.8 °C (>=100.0 °F) (Oral or Oral Equivalent)
Description: For the Concomitant Vaccination group, temperatures were collected after the Day 1 vaccination and the Month 1 visit; for the Non-concomitant Vaccination group, temperatures were collected after the Day 1 vaccination and the Month 1 vaccination.
Time Frame: Up to 5 days following the Day 1 and Month 1 vaccination / visit
Population: The population analyzed included all vaccinated participants with follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 610 | 606
Percentage of participants | 7.7 | 8.1
Statistical Analysis 1: Comparison: Concomitant Vaccination vs Non-concomitant Vaccination; Test type: Superiority or Other; p = 0.806, Miettinen and Nurminen; Difference in percentage = -0.4, 95% CI 2-sided [-3.5 to 2.7]

8. Secondary Outcome: Percentage of Participants Who Seroconvert for Each of the HPV Types Contained in V503
Description: Blood was drawn at Month 7 and assayed to determine whether or not a participant had achieved seroconversion for the HPV types. The lower limit of the titer (milli Merck U/mL) considered seropositive was as follows: HPV Type 6: >=30, HPV Type 11: >=16; HPV Type 16: >=20, HPV Type 18: >=24, HPV Type 31: >=10, HPV Type 33: >=8, HPV Type 45: >=8, HPV Type 52: >=8, and HPV Type 58: >=8.
Time Frame: Month 7
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
Percentage of participants
  Anti-HPV 6: n=501, 514 | 100.0 | 100.0
  Anti-HPV 11: n=502, 514 | 100.0 | 100.0
  Anti-HPV 16: n=513, 530 | 100.0 | 100.0
  Anti-HPV 18: n=516, 535 | 100.0 | 100.0
  Anti-HPV 31: n=514, 536 | 100.0 | 100.0
  Anti-HPV 33: n=520, 537 | 100.0 | 100.0
  Anti-HPV 45: n=523, 539 | 100.0 | 100.0
  Anti-HPV 52: n=521, 538 | 100.0 | 100.0
  Anti-HPV 58: n=519, 537 | 100.0 | 100.0

9. Secondary Outcome: Geometric Mean Titers of the Antibody Response to Neisseria Meningitidis Serogroups Contained in Menactra™
Description: Serum bactericidal antibodies to Neisseria meningitidis serogroups A, C, Y, and W-135 were measured by incubating serial dilutions of serum with target N. meningitidis strains and complement, and enumerating the surviving bacteria after overnight incubation on blood agar plates. The antibody titer is expressed as the reciprocal of the highest dilution that achieves >50% bacterial killing; a higher value represents a greater antibody response. For the Concomitant Vaccination group, serum samples were collected 4 weeks after Day 1 vaccination; for the Non-concomitant Vaccination group, serum samples were collected 4 weeks after Month 1 vaccination.
Time Frame: 4 weeks following Day 1 or Month 1 vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Number analyzed (Participants) | 619 | 618
Titer
  Serogroup A: n=595, 567 | 4832.7 [4499.9 to 5190.0] | 4365.6 [4057.9 to 4696.6]
  Serogroup C: n=595, 567 | 1002.8 [861.7 to 1167.2] | 1068.4 [914.5 to 1248.1]
  Serogroup Y: n=595, 567 | 1416.2 [1230.5 to 1629.9] | 1066.7 [923.6 to 1231.9]
  Serogroup W-135: n=595, 567 | 3998.4 [3474.4 to 4601.5] | 3794.9 [3286.2 to 4382.2]

ADVERSE EVENTS:
Time Frame: Serious adverse events: up to Month 7; Other adverse events: up to Day 15 following any vaccination
Description: Adverse events were collected for all participants who received at least one dose of V503, Menactra™, and Adacel™
Arm/Group | Concomitant Vaccination | Non-concomitant Vaccination
Serious Adverse Events (participants affected / at risk) | 5/613 | 5/611
Other Adverse Events (participants affected / at risk) | 543/613 | 518/611
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=613) | Non-concomitant Vaccination (N=611)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Testicular torsion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concomitant Vaccination (N=613) | Non-concomitant Vaccination (N=611)
Injection-site erythema (General disorders) | 245 (385) | 233 (357)
Injection-site pain (General disorders) | 518 (1373) | 490 (1298)
Injection-site swelling (General disorders) | 276 (492) | 255 (414)
Pyrexia (General disorders) | 88 (111) | 95 (113)
Nasopharyngitis (Infections and infestations) | 32 (36) | 27 (30)
Headache (Nervous system disorders) | 140 (193) | 107 (157)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 32 (34) | 26 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.